CLINICAL TRIAL: NCT06109350
Title: The Effect of Modified Supporting Play, Exploration and Early Development on Motor Performance in Bhutanese Preterm Infants- Randomized Controlled Trial
Brief Title: The Effect of Physical Therapy Intervention on Motor Performance in Bhutanese Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JDWNRH (Other)
Responsible Party: Principal Investigator, Karma Lhaki, Deputy Chief Physiotherapist, JDWNRH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB/Approval/PN/2023/002/564
Record Dates: First submitted 2023-09-21; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double blinded with the outcome assessor blinded to the group allocation and the parent of preterm infants will be blinded since they will be scheduled for appointment on the different day. The outcome assessor will not be disclosed with the infants information, such as age , any medical diagnosis and group identification.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supporting play exploration and early development intervention (Experimental): Preterm infants will receive supporting play exploration and early developmental intervention till 3 months of corrected age.
  Interventions: Other: Supporting play exploration and early developmental intervention(SPEEDI)
- Standard care (Active Comparator): Preterm infants will receive standard care mostly including health education till 3 months of corrected age.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Supporting play exploration and early developmental intervention(SPEEDI) — SPEEDI will be performed by the parents
  Arms: Supporting play exploration and early development intervention
Other: Standard care — Standard care will be performed by the parents
  Arms: Standard care

SUMMARY:
The purpose of this randomized controlled trial is to assess if physical therapy intervention works well to improve motor performance in Bhutanese preterm infants.The main question the study aims to answer is:

Will physical therapy intervention improve the motor performance of preterm infants at 3 months of corrected age when compared to the preterm infants receiving standard care of parental education? In this study the motor performance of the preterm infants receiving physical therapy intervention and standard care will be compared.

DETAILED DESCRIPTION:
After receiving parental consent, preterm infants meeting the eligibility criteria will be enrolled for the study. 28 preterm infants will be enrolled and followed up from 40 weeks till 3 months of corrected age.

The preterm infants in the intervention group will receive modified supporting play, exploration and early development intervention(SPEEDI) and the standard group will receive standard care. The intervention for both groups will be provided by the physical therapists. The SPEEDI intervention should be carried out by the parent for at least 20mins/day for 5 days in a week. The parent will be asked to bring the infants for monthly follow up.

The motor performance of the preterm infants from this two groups will be assessed at 40 weeks, 1, 2 and 3 months of corrected age. The measurement tool that will be used to assess the preterm infants are Test for Infant Motor Performance(TIMP) and Rapid Neurodevelopment Assessment(RNDA). The assessment will be performed by therapist who will be blinded to the group allocation.

The end point of the study is at 3 months of corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 28 -34 weeks of gestation
* Medically stable and off ventilator at the time of discharge from the hospital
* Parents who consent to come for follow up

Exclusion Criteria:

* Cortical blindness or retinopathy of prematurity causing blindness
* Musculoskeletal/congenital abnormalities
* Brain injuries including intra-ventricular hemorrhage (grade 3 and above), hypoxic ischemic encephalopathy and hydrocephalus
* Genetic syndrome
* Family who do not consent
* Parent with physical and psychological problems
* Infants with medical devices such as NG tube and gastrostomy
* Infants who have undergone major surgery

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Compare the motor performance using Test for Infant Motor Performance(TIMP) | 40 weeks, 1, 2, and 3 months of corrected age
  TIMP is a validated tool to measure the motor performance from 34 weeks post menstrual age through 4 months corrected age. The 42 items on the test provides comprehensive assessment of head and trunk control and arms and legs movement. The total score of TIMP ranges from 0-142 with higher scores representing better motor outcome and lower score representing motor delay.

SECONDARY OUTCOMES:
Compare the neurodevelopment using Rapid Neurodevelopment Assessment(RNDA) | 40 weeks, 1, 2, and 3 months of corrected age
  RNDA is a validated tool to assess the neurodevelopment from birth to 2 years. It used to assess developmental domains such as primitive reflex, gross motor, fine motor, vision, hearing, speech, cognition and behavior. The assessment can be interpreted into four categories which are no, mild, moderate and severe impairment.

OTHER OUTCOMES:
Compare the compliance of the parents | 1, 2, and 3 months
  Parental compliance will be measured by the ability of the parent to correctly demonstrate the home program activity when they come for follow up visit .

CONTACTS AND LOCATIONS:
Overall Officials: Karma Lhaki, Principal Investigator — JDWNRH
Locations (1):
- Jigme Dorji Wangchuck National Referral Hospital(JDWNRH), Thimphu, Bhutan

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared after de identification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be maintained securely for at least five years after completion of study and shared.
Access Criteria: To gain access to data, data requestor can email to principal investigator.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT06109350/Prot_SAP_ICF_000.pdf